CLINICAL TRIAL: NCT00008008
Title: CAMP 013:- Tandem Thiotepa Regimen For Selected Malignant Gliomas:1) Primary Or Recurrent Glioblastoma Multiforme (GBM); and 2) Recurrent Anaplastic Astrocytomas (AA), Oligodendrogliomas (O), Oligoastrocytomas (OA), Ependymomas And Primitive Neuroectodermal Tumors (PNET) That Have Either Progressed After Primary Therapy Or Are Refractory To Standard Chemotherapy
Brief Title: Thiotepa Followed by Peripheral Stem Cell or Bone Marrow Transplant in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068362; CPMC-IRB-8017; CPMC-CAMP-013; NCI-G00-1883
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2007-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent adult brain tumor; adult medulloblastoma; adult glioblastoma; adult oligodendroglioma; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult mixed glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; adult giant cell glioblastoma; adult gliosarcoma; adult supratentorial primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Medulloblastoma; Glioblastoma; Oligodendroglioma; Astrocytoma; Ependymoma; Glioma; Familial ependymoma; Gliosarcoma | interventions — Filgrastim; sargramostim; Cyclophosphamide; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: cyclophosphamide
Drug: thiotepa
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy with peripheral stem cell or bone marrow transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase II trial is studying how well thiotepa followed by peripheral stem cell or bone marrow transplant works in treating patients with malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, disease-free interval, and overall survival of patients with malignant glioma treated with high-dose thiotepa followed by autologous peripheral blood stem cell transplantation.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine whether this drug enters the cerebrospinal fluid of these patients.

OUTLINE: Following a course of induction chemotherapy with cyclophosphamide IV over 4 hours, patients receive filgrastim (G-CSF) daily until the completion of peripheral blood stem cell (PBSC) harvesting. PBSCs are collected over 3-5 days. Patients who do not mobilize sufficient cells undergo bone marrow harvest.

Patients receive high-dose thiotepa IV over 5 hours on day -2. PBSCs or bone marrow are reinfused on day 0. Patients receive sargramostim (GM-CSF) subcutaneously daily beginning on day 0 and continuing until blood counts recover. Treatment repeats every 2-3 weeks for a total of 1-4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at every course, then monthly for 6 months, and then every 2 months thereafter.

Patients are followed monthly for 6 months and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 5-40 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Primary or recurrent glioblastoma multiforme (including gliosarcoma) following surgery and radiotherapy or prior conventional chemotherapy (e.g., carmustine or procarbazine, vincristine, and lomustine)
  * Recurrent or refractory anaplastic astrocytoma following any prior therapy (must be chemoresistant)
  * Recurrent or refractory ependymoma or primitive neuroectodermal tumor (PNET) following any prior therapy
  * Recurrent or refractory oligodendroglioma or oligoastrocytoma following any prior therapy (must be chemoresistant)
* Evaluable disease on gadolinium-enhanced MRI
* Ineligible for other high priority national or institutional study (e.g., protocol CAMP-004)

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* LVEF at least 45% by MUGA

Pulmonary:

* DLCO at least 60% of predicted OR
* Approval by pulmonologist

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy
* No concurrent steroids as antiemetics

Radiotherapy:

* See Disease Characteristics
* See Surgery

Surgery:

* See Disease Characteristics
* For patients with glioblastoma multiforme, concurrent surgery and/or stereotactic radiosurgery to reduce tumor bulk allowed

Other:

* No concurrent acetaminophen during chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-09; Primary Completion 2005-06 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Response rate
Disease-free interval
Overall survival
Toxicity

SECONDARY OUTCOMES:
Pharmacokinetics
Presence of high-dose thiotepa in the cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Hesdorffer, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (2):
- United States (2):
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York